CLINICAL TRIAL: NCT01765348
Title: Evaluating Treatment Efficacy of Two Syntactic Treatment Procedures for Children With Specific Language Impairment (SLI): A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, TO Kit Sum, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HKU 753610H; HKU 753610H (Other Grant/Funding Number: Hong Kong General Research Fund)
Record Dates: First submitted 2012-12-23; First posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Language Impairment in School-years
Keywords: language impairment; language disorders; syntax treatment; narrative-based treatment
MeSH Terms: conditions — Language Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sentence combining (Experimental)
  Interventions: Behavioral: Syntax treatment via sentence-combining method
- Narrative based method (Active Comparator)
  Interventions: Behavioral: Syntax treatment managed by narrative-based treatment

INTERVENTIONS:
Behavioral: Syntax treatment via sentence-combining method — Sentence combining method is a discrete trial method that teaches children to form complex sentences of a same structure through drilling and modeling.
  Treatments are conduced by school-speech therapist once two weeks for 8 sessions.
  Arms: Sentence combining
Behavioral: Syntax treatment managed by narrative-based treatment — Target structures are embedded into narrative stories. Children are exposed to these stories and are scaffolded to form the target sentence structure through answering questions, cloze passage and story retell. Treatment are conduced by school-speech therapist once two weeks for 8 sessions.
  Arms: Narrative based method

SUMMARY:
Specific-language-impairment (SLI) is defined as a significant disorder in language development, which affects one's daily functioning, but not attributable to sensory, intellectual or neuropsychological deficit. Children with SLI make up one of the largest subgroups of students with special educational needs (SEN) in Hong Kong. Without appropriate intervention, SLI may persist into adolescence and lead to long-term literacy difficulties and social rejection, which were found to be associated with societal problems like unemployment and crime commitment. Among the language domains, syntax/grammar has been viewed as a core deficit in these children. Speech-Language-Pathologists (SLPs) often provide intervention on this aspect for them. However, very few intervention efficacy studies could be identified.

Without pertinent research evidence, clinical-decision-making in treatment approach selection may be dubious. This study aims to evaluate the efficacy of two procedures for syntax intervention, namely the Sentence-Combining (SC) and Narrative-Based (NAR) procedures using a randomized-controlled-trial (RCT) design. These two procedures have been indicated to be effective in previous case reports and expert opinions. By using the rigorous study design of RCT, this study provides stronger evidence to support clinicians in determining the most effective treatment procedure. To achieve sufficient statistical power to detect the treatment difference, 52 children with SLI will be recruited and randomly assigned to one of the treatment groups. The primary outcome will be measured by a standardized language assessment. Intention-to-treat analysis will be employed. Pre- and post-treatment scores on the outcomes will be subject to analyses of covariance with the pre-treatment scores as the covariate.

ELIGIBILITY:
Inclusion Criteria:

* children in school years who were diagnosed as language with or with speech impairment by a qualified speech therapist; and
* children failed in a standardized language assessment

Exclusion Criteria:

* children with sensory impairment and other diagnosed developmental disorders such as autism.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in language scores based on a standardized language assessment | Children were followed up to 6 months
  All the children were followed for about 6 months in the middle of the school year when they received regular therapy from their school speech-therapists. Children's language skills were assessed by research speech therapists using a standardized language assessment pre and post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carol K. S. To, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Carol K. S. TO, Hong Kong, HK, Hong Kong